CLINICAL TRIAL: NCT00470106
Title: Improving Basic and Social Cognition in Veterans With Schizophrenia
Acronym: IBASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-026-06S
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Schizoaffective Disorder; Schizophrenia
Keywords: Cognition; Remediation; Schizophrenia; Social Cognition
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cognitive Remediation (Active Comparator): cognitive remediation
  Interventions: Behavioral: Cognitive remediation
- Social Cognitive Skills Training (Experimental): social cognitive skills training
  Interventions: Behavioral: Social Cognitive skills training
- Hybrid Intervention (Active Comparator): combined social cognitive and cognitive remediation training
  Interventions: Behavioral: hybrid intervention
- Skills Training (Other): control training
  Interventions: Behavioral: skills training

INTERVENTIONS:
Behavioral: Cognitive remediation — Computer exercises in attention, memory, and speed of processing.
  Arms: Cognitive Remediation
Behavioral: Social Cognitive skills training — Group training on emotion perception, social perception, and understanding others' mental states.
  Arms: Social Cognitive Skills Training
Behavioral: hybrid intervention — A combination of the two groups listed above.
  Arms: Hybrid Intervention
Behavioral: skills training — Skills training in how to identify symptoms of illness and medication side effects.
  Arms: Skills Training

SUMMARY:
Veterans with schizophrenia and schizoaffective disorder experience very high levels of disability and poor community outcome. Further improvements in community outcome for patients with these disorders will not occur simply through better control of clinical symptoms. Instead, it will be necessary to find treatments that address the key determinants of poor functional outcome. Evidence strongly suggests that basic (non-social) cognitive and social cognitive deficits are among the key determinants of functional outcome for these illnesses. The primary goal of this 2-year pilot study is to implement and validate a new remediation program for social cognition that is appropriate for veterans with schizophrenia and schizoaffective disorder.

DETAILED DESCRIPTION:
Veterans with schizophrenia and schizoaffective disorder experience very high levels of disability and poor community outcome. Further improvements in community outcome for patients with these disorders will not occur simply through better control of clinical symptoms. Instead, it will be necessary to find treatments that address the key determinants of poor functional outcome. Evidence strongly suggests that basic (non-social) cognitive and social cognitive deficits are among the key determinants of functional outcome for these illnesses. The primary goal of this 2-year pilot study is to implement and validate a new remediation program for social cognition that is appropriate for veterans with schizophrenia and schizoaffective disorder.

We plan to recruit 72 patients over the 2 years of the study from the outpatient clinics at the VA Greater Los Angeles Healthcare System (VAGLAHS). They will receive baseline assessment that includes measures of social cognition, basic cognition, electrophysiology, functional capacity, clinical symptoms, community status, and demographics / clinical history. Follow up assessments will be administered at the mid-point of training (at 6 weeks) and end of training (at 12 weeks). Each follow up assessment will include measures of basic cognition, social cognition, electrophysiology, functional capacity, and clinical symptoms. The tester administering the assessments will be blind to treatment group.

Subjects will be randomly assigned to one of four groups: 1) social cognitive training, 2) basic cognitive remediation, 3) a combined social cognitive and basic cognitive intervention, or 4) social skills training. All groups will meet in one-hour sessions held twice a week over the course of 12 weeks in small groups of 3-6. The Social Cognition Intervention (SCI) is a new 24-session, manualized intervention program specifically designed to improve emotion perception, social context processing, and theory of mind / attributional bias in veterans with schizophrenia and schizoaffective disorder. The Basic Cognitive Intervention (BCI) will involve computer-assisted training exercises. Each participant will work individually on a notebook computer. The combined intervention will cover the same content areas as the social cognitive and basic cognitive interventions, but will not go into as much detail as the separate intervention programs. The control condition will be facilitated discussion of current events. Treatment will be administered in a group format with three to six patients and a training coach.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be diagnosed with Schizophrenia, Schizoaffective Disorder, or Psychosis not otherwise specified according to Diagnosis and Statistical Manual-IV criteria.
* In addition, the subjects will meet the following criteria:

  * Between 18 and 60 years of age
  * Estimated premorbid intelligence quotient > 70 (based on reading ability)
  * Understand spoken English sufficiently to comprehend testing procedures
  * Clinically stable (e.g., no inpatient hospitalization in the 8 weeks prior to enrollment, no significant changes in medication in the 6 weeks prior to enrollment, and none anticipated for the 3 months of participation)

Exclusion Criteria:

* No clinically significant neurological disease as determined by medical history
* No history of serious head injury (e.g., loss of consciousness longer than 1 hour)
* No physical, cognitive, or language impairment of such severity as to adversely affect the validity of data
* No evidence of drug or alcohol dependence in the past six months, and not intoxicated at time of testing
* The patients psychotic experiences can be explained solely by the use of drugs or alcohol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Green, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Horan WP, Kern RS, Tripp C, Hellemann G, Wynn JK, Bell M, Marder SR, Green MF. Efficacy and specificity of social cognitive skills training for outpatients with psychotic disorders. J Psychiatr Res. 2011 Aug;45(8):1113-22. doi: 10.1016/j.jpsychires.2011.01.015. Epub 2011 Mar 4. PMID 21377168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient clinics at VA Greater Los Angeles Health care system and local mental health facilities. All patients met Diagnostic and Statistical Manual-IV criteria for schizophrenia, schizoaffective disorder, delusional disorder, or psychosis not otherwise specified (not secondary to substance use disorder)
Pre-assignment Details: This is not a drug study so there is no wash out or run in. Participants were excluded if they did not meet diagnostic criteria.
Groups:
- Social Cognition: Social Cognitive remediation: Group training on emotion perception, social perception, and understanding others' mental states.
- Hybrid Group: Half of the sessions were cognitive remediation and half were social cognitive training.
- Control - Social Skills Training: This group was a control for the amount of time in sessions. There was no social cognitive training.
Period: Overall Study
Arm/Group | Social Cognition | Cognitive Remediation | Hybrid Group | Control - Social Skills Training
Started | 19 | 24 | 21 | 21
Completed | 16 | 19 | 14 | 19
Not Completed | 3 | 5 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Cognition | Cognitive Remediation | Hybrid Group | Control - Social Skills Training | Total
Number analyzed (Participants) | 16 | 19 | 14 | 19 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (7.1) | 46.6 (7.4) | 50.4 (10.1) | 45.1 (11.2) | 48.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4 | 8
  Male | 15 | 17 | 13 | 15 | 60
Region of Enrollment [Number; unit: participants]
  United States | 16 | 19 | 14 | 19 | 68
Affect perception [Mean (Standard Deviation); unit: number of correct answers] — This is a performance-based measure (range 0-56, with higher being better) in which subjects identify the emotion depicted in still photographs of faces. Number of correct identifications is the dependent measure.
  number of correct answers | 37.1 (6.1) | 40.6 (8.4) | 38.6 (8.3) | 43.4 (3.7) | 39.8 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Test Scores for Facial Emotion Identification.
Description: This is a test of social cognition that measures the ability to identify the emotion shown in photos of still faces. The construct of interest is facial affect perception. It is an experimental measure and does not have norms or cut-offs. The range of accuracy scores is 0-56 with higher being better.
Time Frame: Assessments for end point (12 weeks).
Measure: Mean (Standard Deviation); unit: number of correct answers
Arm/Group | Social Cognitive Skills Training | Cognitive Remediation | Hybrid Intervention | Skills Training
Number analyzed (Participants) | 16 | 19 | 14 | 19
number of correct answers | 45.5 (8.2) | 41.1 (12.1) | 43.8 (6.7) | 45.1 (5.0)
Statistical Analysis 1: Comparison: Social Cognitive Skills Training vs Cognitive Remediation vs Hybrid Intervention vs Skills Training; Test type: Superiority or Other; p < .001, mixed model — Not corrected for multiple comparisons because it is primary; same analysis as for secondary outcome variable

2. Secondary Outcome: Mean Test Score From a Test of Functional Capacity (Ability to Perform Daily Activities).
Description: This is a role play demonstration test that measures how well someone handles social communication in daily life. The scores reflect overall effectiveness and are the mean number scored across different social situations with a range of 0-5 with higher being better. There are no norms for this test.
Time Frame: Assessments at endpoint (12 weeks).
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Social Cognition | Cognitive Remediation | Hybrid Group | Control - Social Skills Training
Number analyzed (Participants) | 16 | 19 | 14 | 19
number correct | 3.43 (.78) | 3.57 (.74) | 3.35 (1.11) | 3.19 (.86)
Statistical Analysis 1: Comparison: Social Cognition vs Cognitive Remediation vs Hybrid Group vs Control - Social Skills Training; Test type: Superiority or Other; p < .10, mixed model — A priori threshold for significance was P < .05; Same as for the primary variable

ADVERSE EVENTS:
Time Frame: October 2007 to September 2009
Arm/Group | Social Cognition | Cognitive Remediation | Hybrid Group | Control - Social Skills Training
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/24 | 2/21 | 3/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/24 | 1/21 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Social Cognition (N=19) | Cognitive Remediation (N=24) | Hybrid Group (N=21) | Control - Social Skills Training (N=21)
MRSA cellulitis in both hands. (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
5150 hold for suicidal thinking, aggressive behavior and exessive use of alcohol (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
5150 hold for relapse using cocaine and alcohol (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
5150 for threatening to sexually assault a female Veteran (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subject was hospitalized for 8 days due to an inflammed pancreas. (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
5150 hold for aggressive argument with his mother. (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Social Cognition (N=19) | Cognitive Remediation (N=24) | Hybrid Group (N=21) | Control - Social Skills Training (N=21)
ER visit for public intoxication. (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No